CLINICAL TRIAL: NCT05347160
Title: Evaluation Of Different Pulpotomy Agents Used For Treatment Of Immature Molars (Clinical Trial)
Brief Title: Evaluation Of Different Pulpotomy Agents Used For Treatment Of Immature Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: A04080920
Record Dates: First submitted 2022-03-25; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-03

CONDITIONS: Infected Pulp; Root Canal Treatment
Keywords: Pulpotomy; Calcium Hydroxide; Biodentine; Platelet Rich Fibrin; Open apex; Immature root
MeSH Terms: interventions — tricalcium silicate; Calcium Hydroxide

STUDY DESIGN:
Intervention Model Description: Evaluate the effect of different pulpotomy medicaments on permanent molars with immature root clinically and radiographically:
  1. Calcium Hydroxide
  2. Biodentine
  3. Platelet Rich Fibrin
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- calcium hydroxide : group 1 (Experimental): Immature permanent molars with immature root filled by ca(oh)2
  Interventions: Procedure: Biodentine
- biodentine : group 2 (Experimental): clinically and radiographically evaluate BIODENTINE effect on permanent molars with immature root
  Interventions: Procedure: Biodentine
- platelet rich fibrin : group 3 (Experimental): filling of permanent molars with immature root by platelet rich fibrin
  Interventions: Procedure: Biodentine

INTERVENTIONS:
Procedure: Biodentine — using of biodentine , calcium hydroxide and platelet rich fibrin as pulpotomy agents
  Other Names: Platelet Rich Fibrin (PRF); Calcium Hydroxide CA(oh)2

SUMMARY:
The management of permanent teeth with incomplete root development with compromised pulpal integrity presents a unique challenge. The loss of pulpal vitality before the completion of dentin deposition leaves a weak root more prone to fracture as a result of the thin dentinal walls. Every attempt should be made to preserve the vitality of these immature teeth until maturation has occured.

DETAILED DESCRIPTION:
The management of permanent teeth with incomplete root development with compromised pulpal integrity presents a unique challenge. The loss of pulpal vitality before the completion of dentin deposition leaves a weak root more prone to fracture as a result of the thin dentinal walls. Every attempt should be made to preserve the vitality of these immature teeth until maturation has occured. (1)

Pulpotomy is a universally accepted treatment modality for pulp exposures in immature permanent teeth to preserve the vitality of the radicular pulp and to ensure continued root development. (2) Calcium Hydroxide has been the most commonly utilized pulpotomy agent for vital pulp therapy. However, owing to disadvantages such as degradation over time, formation of tunnel defects beneath dentinal bridges and poor sealing , it is slowly losing its popularity as a first choice agent for pulpotomy. (3)

Vital pulp therapy procedures in permanent teeth with incomplete root development have advanced in recent years. Despite Mineral trioxide aggregate has shown promising potential as a pulpotomy agent , it has some drawbacks that include the presence of toxic elements in the material composition (4) , higher cytotoxicity in its freshly mixed state (5)

,high pH during setting (6) , difficult handling characteristics (7) , long setting time (8) , tooth discoloration (9) and high cost. (10)

Consequently, newer calcium silicate-based materials that retain the desirable properties of original MTA but with easier handling and without tooth discoloration have been introduced . Biodentine has several

advantages, as its good sealing ability, adequate compressive strength , a relatively short initial setting time and the promotion of reparative dentin formation with a positive effect on vital pulp cells. (11, 12)

Recently, Regenerative Medicine , especially at the molecular and cellular level has been given great attention towards 'regeneration' instead of 'replacement' approaches. (13) resulting in 'vital pulp therapy' and regenerative endodontics Concepts. (14) In such treatments, clean environment is believed to be a necessity for further success.

Triple Antibiotic Paste (TAP) , is a combination of 3 antibiotics, ciprofloxacin , metronidazole and Minocycline is widely used to achieve a relatively aseptic environment in the radicular space so that the tissue repair and healing can occur. (15)

Promising results have attracted endodontists and general dental practitioners to endodontic regenerative procedures (ERPs). (16) which is considered as a form of a revolution in root canal therapy. (17-19) Now, it has now been taken into account as an alternative method to traditional calcium hydroxide-induced apexogenesis. (20-21)

Recently, the paste used in the regeneration and revascularization protocol. Studies have shown that the paste can eliminate the root canal microorganisms by removing the diverse groups of obligate and facultative gram-positive and gram-negative bacteria , providing an environment for healing. (22,23)

Platelet-rich fibrin (PRF) is a recent innovation in dentistry that has been prepared and used in 2001. (24) It is considered as an autologous healing biomaterial incorporating leukocytes, platelets, and a wide range of key healing proteins in a dense fibrin matrix. (25) PRF serves as a reservoir for the slow continuous release of growth factors that influence and direct the processes of reparative dentinogenesis (26) . Huang et al (27) investigated the effect of PRF on cultured primary dental pulp cells and concluded that PRF can increase dental pulp cell proliferation and differentiation.

Growth factors included in PRF are mitogenic , chemotactic and angiogenic. Therefore, they appear to be critical to the wound-healing process. PRF induces osteoblasts, gingival fibroblasts, and periodontal ligament cells proliferation as a mitogen . Because of growth factors concentrates, PRF promotes wound healing and regeneration which is used in various disciplines of dentistry to repair and regenerate dental and oral tissues. (28-30)

PRF has anti-inflammatory effect and act as an immune regulation mode. It presented as a perfect scaffold in revascularization of immature permanent teeth with necrotic pulps as it enhances cellular proliferation and differentiation. (31,32)

However, there is a limited number of studies reporting on the success of vital pulp therapy for Immature permanent molars. So, the present study will evaluate different pulpotomy modalities used in Immature permanent molars.

ELIGIBILITY:
Inclusion Criteria:

* Apparent healthy and free from any systemic diseases
* child should have restorable carious first permanent molars with immature root

Exclusion Criteria:

* presence of signs and symptoms of pulp degenration
* presence of internal and external root resorption

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage % of patients with Success | Time Frame: 2 years after restoration procedure
  Percentage of Success of treated infected immaature teeth with diffrent agent. Restorations were given the score Alpha for the ideal clinical situation, Bravo for clinically acceptable and Charlie for clinically unacceptable and in need for replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Salwa M Awad, Prof, Study Director — head of pediatric dentistry and public health department
Locations (1):
- Faculty of Dentistry, Al Mansurah, Dakhalia, Egypt

IPD SHARING:
Plan to Share IPD: No